CLINICAL TRIAL: NCT06753331
Title: A Multicenter, Sham-controlled, Randomized Study to Evaluate the Safety, Tolerability, and Clinical Responses Following Stereotactic Intracranial Implantation of DSP-1083 Into Subjects With Parkinson's Disease
Brief Title: A Multicenter Study to Evaluate Safety, Tolerability, and Clinical Responses of DSP-1083 Into Subjects With Parkinson's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DD201101
Record Dates: First submitted 2024-11-19; First posted 2024-12-31 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The sentinel cohort of 3 to 5 subjects will be open-label and receive DSP-1083. Cohort 2 (20 subjects) will be randomized in a 1:1 ratio to receive either DSP-1083 during a surgical procedure, or sham surgery with no DSP-1083 administered.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DSP-1083 (Experimental): Implantation of DSP-1083 (2.7M viable cells per hemisphere; 5.4M total cell dose)
  Interventions: Combination Product: DSP-1083 implantation
- Sham Surgery (Sham Comparator): Sham surgery subjects will undergo a partial thickness burr hole surgical procedure on each side of the skull with no DSP-1083 administration.
  Interventions: Procedure: Sham surgery treatment

INTERVENTIONS:
Combination Product: DSP-1083 implantation — DSP-1083 subjects will receive 2.7M viable cells per hemisphere; 5.4M total cell dose as implants.
  Arms: DSP-1083
Procedure: Sham surgery treatment — Sham surgery subjects will undergo a partial thickness burr hole surgical procedure on each side of the skull with no DSP-1083 administration.
  Arms: Sham Surgery

SUMMARY:
The Goal of this study is to evaluate the safety, tolerability, and clinical responses following implantation of DSP-1083. Study enrolls both male and female patients in 2 cohorts. This study will be held in approximately 5-8 study sites in United States

DETAILED DESCRIPTION:
This is a multicenter first-in-human (FIH) study designed to evaluate the safety, tolerability, and clinical responses following implantation of dopaminergic progenitor cells derived from induced pluripotent stem cells (DSP-1083) compared with sham surgery. Safety is measured based on adverse events, changes in neuropsychiatric/cognition status, and serial neuroimaging (ie, engraftment status, graft expansion, rejection) over 104 weeks.

Cohort 1 sentinel subject (SS1) will undergo 2 unilateral surgical procedures separated by approximately 28 weeks, whereas SS2 and all subsequent subjects will undergo 1 bilateral surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥ 40 and < 70 years at the time of informed consent with a clinically established diagnosis of Parkinson's disease in accordance with the Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Parkinson's Disease.
2. Subject has a clinically established diagnosis of PD for ≥ 4 years.
3. Subject has suboptimal control of PD symptoms, with optimized oral antiparkinsonian medication regimen including levodopa/carbidopa monotherapy or levodopa/carbidopa plus antiparkinsonian medications, with stable dosing for ≥ 2months prior to screening.
4. Subject has a L-DOPA response of ≥ 30% without the influence of antiparkinsonian medications at Screening.
5. Subject has a Modified Hoehn and Yahr stage 3 - 4 in the Off state.
6. Subject has a pretreatment 18F-DOPA PET scan consistent with PD.
7. Subject has both On and Off states as demonstrated by the MDS-UPDRS Part III/IV and the Hauser patient daily diary.
8. Subjects must meet the following race criteria: 2 of the up to 5 sentinel subjects will be of Asian race, defined as having at least 2 grandparents who are Japanese, Taiwanese, Korean, or Chinese. Subjects in Cohort 2 can be of any race.
9. Subject is approved by the Enrollment Authorization Eligibility Committee following review of all required information collected during Screening.

Exclusion Criteria:

1. Subject has a typical parkinsonian syndrome (eg, progressive supranuclear palsy [PSP], multiple system atrophy [MSA], dementia with Lewy bodies [DLB], corticobasal degeneration, Parkinson-plus syndrome, vascular parkinsonism, secondary parkinsonism, hereditary parkinsonism).
2. Subject has non-PD neurological symptoms or evidence of non-PD brain disease (eg, tumor, inflammation, active or history of vascular disorder, history of cerebral hemorrhage, Alzheimer's disease, or other neurodegenerative disorder) based on neuroimaging and/or medical history that would preclude study participation.
3. Subject has psychiatric symptoms, cognitive impairment, depression, dementia, or other behavioral disorder that would preclude study participation based on Investigator decision.
4. Subject has received previous striatal or other extrapyramidal system PD treatments, including deep-brain stimulation, central nervous system (CNS) ablation (eg, pallidotomy, thalamotomy), implanted cell, or gene therapy, and/or focused ultrasound therapy.
5. Subject has peak-dose dyskinesia of sufficient severity that precludes study participation, defined as any item score of ≥ 3 (moderate dyskinesia) on the UDysRS Part 1B (Patient Dyskinesia Questionnaire) AND/OR any item score of ≥ 2 (moderate dyskinesia) on Part 3 (Objective Evaluation of Dyskinesia Disability) Intensity Scale: Impairment. Subject has another type (eg, diphasic dyskinesia) or an unusual pattern of dyskinesia.
6. Subject has a history of, or concurrent abnormal immune function that may adversely affect the engraftment of the cell implants and use of adjunctive immunosuppressants.
7. The subject has the following clinical laboratory test results at Screening:

   * Neutrophil count < 2,000/μL.
   * Platelet count < 5.0 × 104/μL.
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 3.0 × upper limit of normal.
   * Total bilirubin > 1.5 × upper limit of normal.
   * Persistent estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2.
   * Poorly controlled blood glucose in diabetic subjects (glycosylated hemoglobin > 9.0%, or fasting serum glucose ≥ 200mg/dL).
8. Subject has any disorder that would contraindicate general anesthesia, conscious sedation or stereotactic surgery.
9. Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that would pose a risk to the subject or that might confound the results of the study. In cases in which the impact of the condition upon risk to subject or study results is unclear, the Medical Monitor should be consulted.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2030-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events. | Up to 104 weeks
Incidence of Serious Adverse Events (SAE). | Up to 104 weeks
Incidence and severity of Adverse Events of Special Interest (AESI). | Up to 104 weeks
Incidence and severity of Adverse Events leading to study discontinuation. | Up to 104 weeks
Change from baseline in cognition and neuropsychiatric status as assessed by Montreal Cognitive Assessment (MoCA). | Up to 104 weeks
  The MoCA is a widely used, sensitive, validated screening test for detecting mild cognitive impairment and can also predict the presence of cognitive deterioration (ie, progression from mild cognitive impairment to dementia) in PD patients.
Change from baseline in cognition and neuropsychiatric status as assessed by Mattis Dementia Rating Scale (MDRS). | Up to 104 weeks
  The MDRS has been utilized for early detection of dementia, differential diagnosis between Alzheimer's disease and other dementias. The 144-point scale is an aggregate score of 5 subscales: attention, initiation/perseveration (I/P), construction, conceptualization, and memory.The total score ranges from 0 to 144, with lower scores indicating greater cognitive impairment.
Change from baseline in Head Magnetic Resonance Imaging (MRI) (graft expansion/rejection) neuroimaging parameters. | Up to 104 weeks
  Safety MRIs - are conducted to assess the safety of DSP-1083 including rejection, abnormal growth, and formation of mass lesions, which could indicate teratoma formation
Change from baseline in Fluorodopa (F-DOPA) uptake (graft function) neuroimaging parameters. | Up to 104 weeks
  PET scans using F-DOPA will be performed at Screening and then post-surgery to follow the course of graft development and to provide a measure of dopaminergic nerve terminals in the striatum.
Frequency of subjects with suicidal ideation or suicidal behavior using the Columbia Suicide Severity Scale (C-SSRS). | Up to 104 weeks
Observed values and change from baseline in clinical laboratory tests. | Up to 104 weeks
  Laboratory results at each time point will be summarized using descriptive statistics (mean, standard deviation (SD), median, minimum, and maximum) by treatment group.
Observed values and change from baseline in Heart Rate (HR). | Up to 104 weeks
  12-lead ECG parameters ventricular HR at each time point will be summarized by treatment group. All ECG diagnostic findings will be summarized on the basis of incidence rates by treatment group.
Observed values and change from baseline in QT interval. | Up to 104 weeks
  12-lead ECG parameters QT interval at each time point will be summarized by treatment group. All ECG diagnostic findings will be summarized on the basis of incidence rates by treatment group.
Observed values and change from baseline in PR interval. | Up to 104 weeks
  12-lead ECG parameters PR interval at each time point will be summarized by treatment group. All ECG diagnostic findings will be summarized on the basis of incidence rates by treatment group.
Observed values and change from baseline in QRS duration. | Up to 104 weeks
  12-lead ECG parameters QRS duration at each time point will be summarized by treatment group. All ECG diagnostic findings will be summarized on the basis of incidence rates by treatment group.
Observed values and change from baseline in RR interval. | Up to 104 weeks
  12-lead ECG parameters RR interval at each time point will be summarized by treatment group. All ECG diagnostic findings will be summarized on the basis of incidence rates by treatment group.
Observed values and change from baseline in QTcF interval. | Up to 104 weeks
  12-lead ECG parameters QTcF interval at each time point will be summarized by treatment group. All ECG diagnostic findings will be summarized on the basis of incidence rates by treatment group.
Observed values and change from baseline in body temperature. | Up to 104 weeks
  Vital signs parameter body temperature will be summarized using descriptive statistics at each time point by treatment group.
Observed values and change from baseline in respiratory rate. | Up to 104 weeks
  Vital signs parameter supine respiratory rate will be summarized using descriptive statistics at each time point by treatment group.
Observed values and change from baseline in pulse rate. | Up to 104 weeks
  Vital signs parameter supine and standing pulse will be summarized using descriptive statistics at each time point by treatment group.
Observed values and change from baseline in Systolic Blood Pressure. | Up to 104 weeks
  Vital signs parameter Systolic Blood Pressure will be summarized using descriptive statistics at each time point by treatment group.
Observed values and change from baseline in Diastolic Blood Pressure. | Up to 104 weeks
  Vital signs parameter Diastolic Blood Pressure will be summarized using descriptive statistics at each time point by treatment group.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kentucky Medical Center, Lexington, Kentucky
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York